CLINICAL TRIAL: NCT01478217
Title: Positive End-expiratory Pressure Induced Lung Recruitment -Comparison Between Ultrasonographic Assessment and Lower Inflection Point Assessment on the Pressure -Volume Loop
Brief Title: PEEP Recruitment-comparison Between Ultrasonographic Assessment and LIP Assessment
Status: Completed | Type: Observational
Sponsor: Sisters of Mercy University Hospital (Other)
Responsible Party: Principal Investigator, Bojan Rode, dr.med., Sisters of Mercy University Hospital
Other Study IDs: Vinogradska29
Record Dates: First submitted 2011-11-20; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: lung ultrasonography; pressure-volume loops; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare lung recruitment in acute lung injury (ALI)/acute respiratory distress syndrome (ARDS) based on lower inflection point with transthoracic ultrasonographic assessment of lung recruitment.

DETAILED DESCRIPTION:
Sedated and sometimes temporary relaxed patients with ALI/ARDS on mechanical ventilation in semirecumbent position are included. Lower inflection point on pressure volume loop on ventilator Draeger Evita 4 with low continuous flow on volume controlled ventilation is measured with zero PEEP. Transthoracic lung ultrasound with linear probe is proceed on both hemithoraces when mechanical ventilation based on measured PEEP is started. We compare if real lung recruitment seen by ultrasound is the same as predicted by lower inflection point.

The procedure is a part of routine everyday respiratory monitoring in our unit.

ELIGIBILITY:
Inclusion Criteria:

* patients with diffuse ALI/ARDS on mechanical ventilation with visible lower inflection point on dynamic P-V loops

Exclusion Criteria:

* preexisting parenchymal or pleural lung disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Rode, M.D., Principal Investigator
Locations (1):
- Central intensive care unit, University hospital "Sisters of Mercy", Grad Zagreb, Croatia

REFERENCES:
- [Result] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923